CLINICAL TRIAL: NCT03391986
Title: Auricular Acupuncture as Adjunct for Pain Management During First Trimester Uterine Aspiration.
Brief Title: Acupuncture for Pain Management During Uterine Aspiration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Society of Family Planning (Other)
Responsible Party: Principal Investigator, Carolyn Westhoff, Professor of Epidemiology and Population and Family Health, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: AAAR2610
Record Dates: First submitted 2017-11-06; First posted 2018-01-05 (Actual); Results first posted 2019-09-03 (Actual); Last update posted 2019-09-03 (Actual); Status verified 2019-08

CONDITIONS: Pain Acute; Acupuncture
MeSH Terms: conditions — Acute Pain | interventions — Needles; Acupuncture Therapy

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to either 1 - auricular acupuncture with pyonex needle, 2 - placebo adhesive, or 3 - routine care using a 1:1:1 ratio. The randomization scheme will use randomly permuted blocks with a block size of 6 or 9.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participant: only participants in the pyonex needle and placebo adhesive group will be masked during the study. Equipment is opened behind the participant and the needles and adhesives are placed outside the view of the participant.
  Care Provider: A colored hat that covers the participants ears will be placed. Outcomes Assessor: Group assignment will be masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Pyonex needles (Active Comparator): This arm will receive modified battlefield auricular acupuncture using SEIRIN® Pyonex™ Acupuncture Needles.
  Interventions: Device: SEIRIN® Pyonex™ Acupuncture Needles
- Placebo adhesives (Placebo Comparator): This arm will receive placement of adhesives using the modified battlefield auricular acupuncture placement points using 12 mm Plasters.
  Interventions: Procedure: 12 mm Plasters
- Routine Care (No Intervention): This arm will receive no intervention.

INTERVENTIONS:
Device: SEIRIN® Pyonex™ Acupuncture Needles — Needles will be placed on the right and left ear. Right ear - cingulate gyrus, thalamus, Point Zero, Shen Men, uterus. Left ear - cingulate gyrus, thalamus, Point Zero, Shen Men, cervix
  Other Names: Needle, Acupuncture, Single Use
  Arms: Pyonex needles
Procedure: 12 mm Plasters — 12 mm (0.5"). Latex-free Adhesives will be placed on the right and left ear. Right ear - cingulate gyrus, thalamus, Point Zero, Shen Men, uterus. Left ear - cingulate gyrus, thalamus, Point Zero, Shen Men, cervix
  Other Names: hypoallergenic, adhesive replacement plasters
  Arms: Placebo adhesives

SUMMARY:
The proposed study will be a randomized, double blinded, placebo-controlled trial to evaluate the efficacy of auricular acupuncture as adjunct for pain management during abortion. Women seeking first trimester uterine aspiration procedure who enroll in the study will be randomized to receive: 1) auricular acupuncture using pyonex needles, 2) placebo using an adhesive, 3) or routine care. Both participants and the treating physician will be unaware of treatment assignment. The primary outcome will compare the maximum pain score as measured by the visual analog scale (VAS) between the auricular acupuncture group and the routine care group. The secondary outcome will compare the maximum pain score between placebo group to the routine care group. The study will also investigate patient satisfaction.

DETAILED DESCRIPTION:
Of the estimated 1.06 million abortions performed in the United States in 2011, approximately 91% occurred before 13 weeks gestation. Most first trimester abortions are performed in an outpatient center with a paracervical block as the only analgesic. Paracervical block is associated with improved pain control during dilation and aspiration however, women still experience moderate to severe pain. Moderate sedation and general anesthesia, minimize pain more than a paracervical block; however increased cost, regulatory constraints, side effects, health risks, and recovery time may limit abortion access.

Pain experienced during abortion results from a complex interaction of physical innervation pathways, psychological and social factors. Pain during abortion is also influenced by additional factors such as age, pregnancy history, and self-reported pre-procedure anxiety about abortion. Adequate pain management during suction aspiration might require interventions that influence mental and emotional states as well as physical pain.

Acupuncture affects perception of painful stimuli and improves anxiety. Peripheral stimulation of acupoints mobilizes central neuropeptides involved in the pathway of anxiety and stress. In auricular acupuncture, a technique of acupuncture, needles are placed in designated acupoints on the external ear in order to alleviate health conditions, in particular pain, in other parts of the body.

In a pilot study completed at Columbia University Medical Center (CUMC) in 2016, patients seeking first trimester uterine aspiration were interested in the complementary medicine technique of auricular acupuncture as an adjunct to local anesthesia. Currently, the effectiveness of auricular acupuncture to control pain during a uterine suction aspiration is unknown.

Participants will be randomized to either auricular acupuncture with pyonex needle adhesives, placebo adhesive, or routine care using a 1:1:1 ratio. The randomization scheme will use randomly permuted blocks with a block size of 4 or 6. An investigator experienced with generating randomization sequences and not directly involved in the study will be responsible for creating the entire randomized schedule; first by defining the sequence of block sizes and second, by defining the assignments within each block. The division research office at CUMC will prepare opaque, sealed envelopes containing cards indicating whether a given patient has been randomized to receive either pyonex needles, placebo adhesive, or routine care. The allocation will remain concealed from the patient and abortion provider. The acupuncturist will open the sealed, opaque envelope immediately prior to the suction aspiration procedure and perform the intervention according to randomization assignment.

ELIGIBILITY:
Inclusion Criteria:

* English- or Spanish-speaking women
* Age 18 or older
* Seeking first trimester suction aspiration for undesired pregnancy, early pregnancy failure, retained products of conception, or molar pregnancy
* Intrauterine pregnancy with gestational age less than or equal to 12 weeks and 6 days
* Willingness to receive acupuncture and be randomized in the study

Exclusion Criteria:

* Allergy to adhesives
* Allergy to or cannot receive ibuprofen or 1% lidocaine
* Congenital anomalies of the ear including anotia and microtia

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 153 (Actual)
Dates: Start 2017-09-09 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Westhoff, MD MSc, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Allen RH, Fitzmaurice G, Lifford KL, Lasic M, Goldberg AB. Oral compared with intravenous sedation for first-trimester surgical abortion: a randomized controlled trial. Obstet Gynecol. 2009 Feb;113(2 Pt 1):276-83. doi: 10.1097/AOG.0b013e3181938758. PMID 19155895
- [Background] Allen RH, Kumar D, Fitzmaurice G, Lifford KL, Goldberg AB. Pain management of first-trimester surgical abortion: effects of selection of local anesthesia with and without lorazepam or intravenous sedation. Contraception. 2006 Nov;74(5):407-13. doi: 10.1016/j.contraception.2006.06.002. Epub 2006 Aug 2. PMID 17046383
- [Background] Allen RH, Micks E, Edelman A. Pain relief for obstetric and gynecologic ambulatory procedures. Obstet Gynecol Clin North Am. 2013 Dec;40(4):625-45. doi: 10.1016/j.ogc.2013.08.005. PMID 24286993
- [Background] Bae H, Bae H, Min BI, Cho S. Efficacy of acupuncture in reducing preoperative anxiety: a meta-analysis. Evid Based Complement Alternat Med. 2014;2014:850367. doi: 10.1155/2014/850367. Epub 2014 Sep 2. PMID 25254059
- [Background] Belanger E, Melzack R, Lauzon P. Pain of first-trimester abortion: a study of psychosocial and medical predictors. Pain. 1989 Mar;36(3):339-350. doi: 10.1016/0304-3959(89)90094-8. PMID 2710563
- [Background] Borup L, Wurlitzer W, Hedegaard M, Kesmodel US, Hvidman L. Acupuncture as pain relief during delivery: a randomized controlled trial. Birth. 2009 Mar;36(1):5-12. doi: 10.1111/j.1523-536X.2008.00290.x. PMID 19278378
- [Background] Chan AW, Tetzlaff JM, Altman DG, Laupacis A, Gotzsche PC, Krleza-Jeric K, Hrobjartsson A, Mann H, Dickersin K, Berlin JA, Dore CJ, Parulekar WR, Summerskill WS, Groves T, Schulz KF, Sox HC, Rockhold FW, Rennie D, Moher D. SPIRIT 2013 statement: defining standard protocol items for clinical trials. Ann Intern Med. 2013 Feb 5;158(3):200-7. doi: 10.7326/0003-4819-158-3-201302050-00583. PMID 23295957
- [Background] Eghbali M, Yekaninejad MS, Varaei S, Jalalinia SF, Samimi MA, Sa'atchi K. The effect of auricular acupressure on nausea and vomiting caused by chemotherapy among breast cancer patients. Complement Ther Clin Pract. 2016 Aug;24:189-94. doi: 10.1016/j.ctcp.2016.06.006. Epub 2016 Jul 5. PMID 27502820
- [Background] Ekdahl L, Petersson K. Acupuncture treatment of pregnant women with low back and pelvic pain--an intervention study. Scand J Caring Sci. 2010 Mar;24(1):175-82. doi: 10.1111/j.1471-6712.2009.00704.x. Epub 2010 Jan 20. PMID 20102541
- [Background] Facco E, Stellini E, Bacci C, Manani G, Pavan C, Cavallin F, Zanette G. Validation of visual analogue scale for anxiety (VAS-A) in preanesthesia evaluation. Minerva Anestesiol. 2013 Dec;79(12):1389-95. Epub 2013 Jul 9. PMID 23860442
- [Background] Feng X, Ye T, Wang Z, Chen X, Cong W, Chen Y, Chen P, Chen C, Shi B, Xie W. Transcutaneous acupoint electrical stimulation pain management after surgical abortion: A cohort study. Int J Surg. 2016 Jun;30:104-8. doi: 10.1016/j.ijsu.2016.04.042. Epub 2016 Apr 29. PMID 27142864
- [Background] Frye LJ, Chong E, Winikoff B; NCT01799252 Trial Investigators. What happens when we routinely give doxycycline to medical abortion patients? Contraception. 2015 Jan;91(1):19-24. doi: 10.1016/j.contraception.2014.09.001. Epub 2014 Sep 15. PMID 25444253
- [Background] Guerrero JM, Castano PM, Schmidt EO, Rosario L, Westhoff CL. Music as an auxiliary analgesic during first trimester surgical abortion: a randomized controlled trial. Contraception. 2012 Aug;86(2):157-62. doi: 10.1016/j.contraception.2011.11.017. Epub 2012 Jan 10. PMID 22240180
- [Background] Holzer A, Leitgeb U, Spacek A, Wenzl R, Herkner H, Kettner S. Auricular acupuncture for postoperative pain after gynecological surgery: a randomized controlled trail. Minerva Anestesiol. 2011 Mar;77(3):298-304. PMID 21441884
- [Background] Jamison RN, Gracely RH, Raymond SA, Levine JG, Marino B, Herrmann TJ, Daly M, Fram D, Katz NP. Comparative study of electronic vs. paper VAS ratings: a randomized, crossover trial using healthy volunteers. Pain. 2002 Sep;99(1-2):341-7. doi: 10.1016/s0304-3959(02)00178-1. PMID 12237213
- [Background] Jensen MP, Miller L, Fisher LD. Assessment of pain during medical procedures: a comparison of three scales. Clin J Pain. 1998 Dec;14(4):343-9. doi: 10.1097/00002508-199812000-00012. PMID 9874014
- [Background] Jensen MP, Chen C, Brugger AM. Interpretation of visual analog scale ratings and change scores: a reanalysis of two clinical trials of postoperative pain. J Pain. 2003 Sep;4(7):407-14. doi: 10.1016/s1526-5900(03)00716-8. PMID 14622683
- [Background] Jones RK, Jerman J. Abortion incidence and service availability in the United States, 2011. Perspect Sex Reprod Health. 2014 Mar;46(1):3-14. doi: 10.1363/46e0414. Epub 2014 Feb 3. PMID 24494995
- [Background] Kindberg S, Klunder L, Strom J, Henriksen TB. Ear acupuncture or local anaesthetics as pain relief during postpartum surgical repair: a randomised controlled trial. BJOG. 2009 Mar;116(4):569-76. doi: 10.1111/j.1471-0528.2008.02016.x. Epub 2008 Dec 19. PMID 19120322
- [Background] Kiran G, Gumusalan Y, Ekerbicer HC, Kiran H, Coskun A, Arikan DC. A randomized pilot study of acupuncture treatment for primary dysmenorrhea. Eur J Obstet Gynecol Reprod Biol. 2013 Jul;169(2):292-5. doi: 10.1016/j.ejogrb.2013.02.016. Epub 2013 Mar 20. PMID 23522721
- [Background] Lanser P, Gesell S. Pain management: the fifth vital sign. Healthc Benchmarks. 2001 Jun;8(6):68-70, 62. PMID 11474948
- [Background] Leggit JC. Introduction of Integrative Health and Acupuncture to Pre-Clerkship Medical Students. Med Acupunct. 2014 Aug 1;26(4):226-229. doi: 10.1089/acu.2014.1045. PMID 25184015
- [Background] Micks EA, Edelman AB, Renner RM, Fu R, Lambert WE, Bednarek PH, Nichols MD, Beckley EH, Jensen JT. Hydrocodone-acetaminophen for pain control in first-trimester surgical abortion: a randomized controlled trial. Obstet Gynecol. 2012 Nov;120(5):1060-9. doi: 10.1097/aog.0b013e31826c32f0. PMID 23090523
- [Background] Michalek-Sauberer A, Gusenleitner E, Gleiss A, Tepper G, Deusch E. Auricular acupuncture effectively reduces state anxiety before dental treatment--a randomised controlled trial. Clin Oral Investig. 2012 Dec;16(6):1517-22. doi: 10.1007/s00784-011-0662-4. Epub 2012 Jan 6. PMID 22219023
- [Background] Miyazaki S, Hagihara A, Kanda R, Mukaino Y, Nobutomo K. Applicability of press needles to a double-blind trial: a randomized, double-blind, placebo-controlled trial. Clin J Pain. 2009 Jun;25(5):438-44. doi: 10.1097/AJP.0b013e318193a6e1. PMID 19454879
- [Background] O'Connell K, Jones HE, Simon M, Saporta V, Paul M, Lichtenberg ES; National Abortion Federation Members. First-trimester surgical abortion practices: a survey of National Abortion Federation members. Contraception. 2009 May;79(5):385-92. doi: 10.1016/j.contraception.2008.11.005. Epub 2008 Dec 11. PMID 19341852
- [Background] Oleson, T (1998). "Auriculotherapy Manual: Chinese and Western Systems of Ear Acupuncture, 2nd edition." California, Health Care Alternatives, Inc
- [Background] Pazol K, Creanga AA, Burley KD, Jamieson DJ. Abortion surveillance - United States, 2011. MMWR Surveill Summ. 2014 Nov 28;63(11):1-41. PMID 25426741
- [Background] Platon B, Andrell P, Raner C, Rudolph M, Dvoretsky A, Mannheimer C. High-frequency, high-intensity transcutaneous electrical nerve stimulation as treatment of pain after surgical abortion. Pain. 2010 Jan;148(1):114-119. doi: 10.1016/j.pain.2009.10.023. Epub 2009 Dec 2. PMID 19959293
- [Background] Renner RM, Jensen JT, Nichols MD, Edelman AB. Pain control in first-trimester surgical abortion: a systematic review of randomized controlled trials. Contraception. 2010 May;81(5):372-88. doi: 10.1016/j.contraception.2009.12.008. Epub 2010 Jan 27. PMID 20399943
- [Background] Renner RM, Edelman AB, Nichols MD, Jensen JT, Lim JY, Bednarek PH. Refining paracervical block techniques for pain control in first trimester surgical abortion: a randomized controlled noninferiority trial. Contraception. 2016 Nov;94(5):461-466. doi: 10.1016/j.contraception.2016.05.005. Epub 2016 May 25. PMID 27235677
- [Background] Rowbotham MC. What is a "clinically meaningful" reduction in pain? Pain. 2001 Nov;94(2):131-132. doi: 10.1016/S0304-3959(01)00371-2. No abstract available. PMID 11690725
- [Background] Schlaeger JM, Gabzdyl EM, Bussell JL, Takakura N, Yajima H, Takayama M, Wilkie DJ. Acupuncture and Acupressure in Labor. J Midwifery Womens Health. 2017 Jan;62(1):12-28. doi: 10.1111/jmwh.12545. Epub 2016 Dec 21. PMID 28002621
- [Background] Shapiro AG, Cohen H. Auxiliary pain relief during suction curettage. Contraception. 1975 Jan;11(1):25-30. doi: 10.1016/0010-7824(75)90047-5. No abstract available. PMID 1116357
- [Background] Smith CA, Crowther CA, Petrucco O, Beilby J, Dent H. Acupuncture to treat primary dysmenorrhea in women: a randomized controlled trial. Evid Based Complement Alternat Med. 2011;2011:612464. doi: 10.1093/ecam/nep239. Epub 2011 Mar 20. PMID 21799683
- [Background] Smith GM, Stubblefield PG, Chirchirillo L, McCarthy MJ. Pain of first-trimester abortion: its quantification and relations with other variables. Am J Obstet Gynecol. 1979 Mar 1;133(5):489-98. doi: 10.1016/0002-9378(79)90282-5. PMID 443287
- [Background] Tangsiriwatthana T, Sangkomkamhang US, Lumbiganon P, Laopaiboon M. Paracervical local anaesthesia for cervical dilatation and uterine intervention. Cochrane Database Syst Rev. 2013 Sep 30;2013(9):CD005056. doi: 10.1002/14651858.CD005056.pub3. PMID 24085642
- [Background] Todd KH, Funk KG, Funk JP, Bonacci R. Clinical significance of reported changes in pain severity. Ann Emerg Med. 1996 Apr;27(4):485-9. doi: 10.1016/s0196-0644(96)70238-x. PMID 8604867
- [Background] Tsai SL, Fox LM, Murakami M, Tsung JW. Auricular Acupuncture in Emergency Department Treatment of Acute Pain. Ann Emerg Med. 2016 Nov;68(5):583-585. doi: 10.1016/j.annemergmed.2016.05.006. Epub 2016 Jun 8. PMID 27287548
- [Background] White K, Jones H, Lichtenberg S, Paul M (2015). "First trimester surgical abortion practices in the United States." Poster presented at: Society of Family Planning Forum in 2015.
- [Background] Wang SM, Dezinno P, Lin EC, Lin H, Yue JJ, Berman MR, Braveman F, Kain ZN. Auricular acupuncture as a treatment for pregnant women who have low back and posterior pelvic pain: a pilot study. Am J Obstet Gynecol. 2009 Sep;201(3):271.e1-9. doi: 10.1016/j.ajog.2009.04.028. Epub 2009 Jun 26. PMID 19560110
- [Background] Wu J, Chaplin W, Amico J, Butler M, Ojie MJ, Hennedy D, Clemow L. Music for surgical abortion care study: a randomized controlled pilot study. Contraception. 2012 May;85(5):496-502. doi: 10.1016/j.contraception.2011.09.018. Epub 2011 Nov 12. PMID 22079604
- [Background] Yeh CH, Chiang YC, Hoffman SL, Liang Z, Klem ML, Tam WW, Chien LC, Suen LK. Efficacy of auricular therapy for pain management: a systematic review and meta-analysis. Evid Based Complement Alternat Med. 2014;2014:934670. doi: 10.1155/2014/934670. Epub 2014 Jul 23. PMID 25165482
- [Background] Zane S, Creanga AA, Berg CJ, Pazol K, Suchdev DB, Jamieson DJ, Callaghan WM. Abortion-Related Mortality in the United States: 1998-2010. Obstet Gynecol. 2015 Aug;126(2):258-265. doi: 10.1097/AOG.0000000000000945. PMID 26241413
- [Result] Ndubisi C, Danvers A, Gold MA, Morrow L, Westhoff CL. Auricular acupuncture as an adjunct for pain management during first trimester abortion: a randomized, double-blinded, three arm trial. Contraception. 2019 Mar;99(3):143-147. doi: 10.1016/j.contraception.2018.11.016. Epub 2018 Dec 7. PMID 30529393
- See also: Guttmacher Institute. 2016. Induced Abortion in the United States — http://www.guttmacher.org/fact-sheet/induced-abortion-united-states

RESULTS

PARTICIPANT FLOW:
Groups:
- Pyonex Needles: This arm will receive modified battlefield auricular acupuncture using SEIRIN® Pyonex™ Acupuncture Needles.
  SEIRIN® Pyonex™ Acupuncture Needles: Needles will be placed on the right and left ear.
  Right ear - cingulate gyrus, thalamus, Point Zero, Shen Men, uterus. Left ear - cingulate gyrus, thalamus, Point Zero, Shen Men, cervix
Period: Overall Study
Arm/Group | Pyonex Needles | Placebo Adhesives | Routine Care
Started | 53 | 50 | 50
Completed | 53 | 50 | 50
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pyonex Needles | Placebo Adhesives | Routine Care | Total
Number analyzed (Participants) | 53 | 50 | 50 | 153
Age, Customized [Mean (Standard Deviation); unit: years]
  Age | 31 (6.8) | 28.7 (6.9) | 30.9 (7.6) | 30.2 (7.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 50 | 50 | 153
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 43 | 39 | 39 | 121
  Not Hispanic or Latino | 7 | 9 | 9 | 25
  Unknown or Not Reported | 3 | 2 | 2 | 7
Region of Enrollment [Number; unit: participants]
  United States | 53 | 50 | 50 | 153
Pregnancy type [Count of Participants; unit: Participants]
  Induced abortion | 39 | 34 | 33 | 106
  Spontaneous abortion | 14 | 16 | 17 | 47

OUTCOME MEASURES:

1. Primary Outcome: Visual Analog Scale for Pain (VAS Pain) Score - Acupuncture Versus Routine Care
Description: Measure effectiveness of auricular acupuncture as an adjunct to ibuprofen and paracervical block for pain control during first trimester uterine aspiration by comparing the maximum pain score; as measured by VAS between women randomized to receive auricular acupuncture and routine care controls - using a 100 mm visual analog scale (VAS-P) (anchors: 0 mm = no pain, 100 mm = worst pain in my life). The VAS has no sub-scales.
Time Frame: at the completion of the procedure (approximately 10 minutes later)
Population: The final analysis included 150 (out of 153) participants: 52 in the auricular acupuncture group, 49 in the placebo group and 49 in the routine (usual) care group.
Measure: Mean (Inter-Quartile Range); unit: score on a scale
Arm/Group | Pyonex Needles | Routine Care
Number analyzed (Participants) | 52 | 49
score on a scale | 39.5 [11 to 63] | 71.0 [33 to 90]

2. Secondary Outcome: Change in Visual Analog Scale for Pain (VAS Pain) Score - Placebo Versus Routine Care
Description: Measure effectiveness of placebo as an adjunct to ibuprofen and paracervical block for pain control during uterine aspiration by comparing the maximum pain score; as measured by VAS between women randomized to receive placebo adhesives and routine care controls - using a 100 mm visual analog scale (VAS-P) (anchors: 0 mm = no pain, 100 mm = worst pain in my life).
Time Frame: prior to the procedure (baseline), at the completion of the procedure (approximately 10 minutes later)
Population: as for outcome 1
Measure: Mean (Inter-Quartile Range); unit: score on a scale
Arm/Group | Placebo Adhesives | Routine Care
Number analyzed (Participants) | 49 | 49
score on a scale | 70.0 [1 to 81] | 71.0 [33 to 90]

3. Secondary Outcome: Percentage of Patients Rated Good or Very Good on Satisfaction Survey in Overall Care - Acupuncture Versus Routine Care
Description: Using a satisfaction survey (investigator-developed, 6 questions, each question is graded on a scale of 1-5, 1 being very poor and 5 being very good) to measure effectiveness of auricular acupuncture for improving satisfaction.
Time Frame: at the completion of the procedure (approximately 5-10 minutes)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Pyonex Needles | Routine Care
Number analyzed (Participants) | 52 | 49
percentage of participants | 94 | 76

ADVERSE EVENTS:
Time Frame: The duration of the procedure (approximately 5-10 minutes)
Arm/Group | Pyonex Needles | Placebo Adhesives | Routine Care
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/49 | 0/49
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/49 | 0/49
Other Adverse Events (participants affected / at risk) | 0/52 | 0/49 | 0/49

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-17): https://cdn.clinicaltrials.gov/large-docs/86/NCT03391986/Prot_SAP_000.pdf